CLINICAL TRIAL: NCT05802238
Title: Efficacy of Tranexamic Acid (TXA) in Humerus ORIF
Acronym: TXA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of staffing
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Peter Tang, Associate Professor of Orthopaedic Surgery, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-153
Record Dates: First submitted 2023-02-08; First posted 2023-04-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-06

CONDITIONS: Fracture Humerus
Keywords: Open Reduction Internal Fixation; Blood loss
MeSH Terms: conditions — Humeral Fractures; Hemorrhage | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Single-center randomized controlled trial, parallel two-arm design allocation 1:1 exposed-control design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Patients randomized to treatment arm of study will have TXA administered 10 minutes prior to surgery
  Interventions: Drug: Tranexamic acid (TXA)
- Control Group (Placebo Comparator): The control group will have saline administered 10 minutes prior to surgery.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Tranexamic acid (TXA) — 1 gram of TXA in 10mg single-dose ampule (100mg/mL) administered 10 minutes prior to surgery
  Other Names: Tranexamic acid
  Arms: Treatment Arm
Other: Saline — control group will receive 10 mL of normal saline infused intravenously at 1 mL/min.
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine if administration of tranexamic acid (TXA), a clotting agent, will decrease blood loss, the need for transfusion, and reduce the likelihood of wound complications such as infection. Investigators will also see if the drug can effectively decrease operative time and length of hospitalization.

DETAILED DESCRIPTION:
Single-center randomized controlled trial, parallel two-arm design allocation 1:1 exposed-control design to determine if TXA aids in prevention of blood loss in upper extremity trauma, specifically humerus fractures. Patient population includes male and female adults with no history of thromboses who suffered an isolated humeral injury. Patients will be evaluated at Allegheny General Hospital (AGH) as surgical candidates and allocated to the exposure group (receive TXA) or the control group (saline placebo). Patients randomized to treatment arm of study will have TXA administered 10 minutes prior to surgery. The control group will have saline administered 10 minutes prior to surgery. Patients will be seen in follow up at both 2 weeks and 6 weeks postoperatively, as well as followed through the electronic medical record (EMR).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 18-100 years
2. Isolated proximal humerus or humeral shaft fracture undergoing open reduction internal fixation.
3. Must be able to read and understand English and consent for themselves.

Exclusion Criteria:

1. Allergy to TXA.
2. Acquired disturbances of color vision.
3. History of arterial or venous thromboembolic disease; such as DVT, PE, CVA, TIA.
4. Pregnant or breastfeeding.
5. Recent MI (within 6 months of surgery) or any placement of stent regardless of time since placement.
6. Renal impairment (creatinine above 1.2 in women, creatinine above 1.4 in men)
7. Refusal of blood products
8. Subarachnoid hemorrhage
9. Disseminated intravascular coagulation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Blood loss | Intraoperatively
  The estimated total blood loss measured intraoperatively. This will be done by estimating absorbed drainage by surgical gauze and adding this to total volume in suction canister. Total volume of irrigation used will be subtracted from this total to give an estimate of intraoperative blood loss.

SECONDARY OUTCOMES:
Operative Time | From the start of surgical procedure through the completion of the surgical procedure
  Amount of time of operative procedure
Duration of follow-up | Through study completion, an average of one year.
  Through study completion, an average of one year.
Complications (DVT, PE, stroke) | through study completion, an average of one year
  Presence or absence of the monitored complications (DVT, PE, stroke) will be recorded as a categorical data value.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tang, MD, Principal Investigator — Allegheny Health Network Allegheny General Hospital
Locations (1):
- Allegheny Health Network Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Arnould G, Hartemann P, Tridon P, Weber M, Floquet J, Cagniart MJ. [Balo's concentric sclerosis with dementia]. Rev Neurol (Paris). 1970 Mar;122(3):203-8. No abstract available. French. PMID 5459718
- [Background] Hughes JM, Seale JP, Temple DM. Effect of fenoterol on immunological release of leukotrienes and histamine from human lung in vitro: selective antagonism by beta-adrenoceptor antagonists. Eur J Pharmacol. 1983 Nov 25;95(3-4):239-45. doi: 10.1016/0014-2999(83)90640-4. PMID 6197312
- [Background] Cheriyan T, Maier SP 2nd, Bianco K, Slobodyanyuk K, Rattenni RN, Lafage V, Schwab FJ, Lonner BS, Errico TJ. Efficacy of tranexamic acid on surgical bleeding in spine surgery: a meta-analysis. Spine J. 2015 Apr 1;15(4):752-61. doi: 10.1016/j.spinee.2015.01.013. Epub 2015 Jan 21. PMID 25617507
- [Background] Yu X, Wang J, Wang X, Xie L, Chen C, Zheng W. The efficacy and safety of tranexamic acid in the treatment of intertrochanteric fracture: an updated meta-analysis of 11 randomized controlled trials. J Thromb Thrombolysis. 2020 Aug;50(2):243-257. doi: 10.1007/s11239-019-02034-1. PMID 31902124
- [Background] Spitler CA, Row ER, Gardner WE 2nd, Swafford RE, Hankins MJ, Nowotarski PJ, Kiner DW. Tranexamic Acid Use in Open Reduction and Internal Fixation of Fractures of the Pelvis, Acetabulum, and Proximal Femur: A Randomized Controlled Trial. J Orthop Trauma. 2019 Aug;33(8):371-376. doi: 10.1097/BOT.0000000000001480. PMID 30939507
- [Background] Baskaran D, Rahman S, Salmasi Y, Froghi S, Berber O, George M. Effect of tranexamic acid use on blood loss and thromboembolic risk in hip fracture surgery: systematic review and meta-analysis. Hip Int. 2018 Jan;28(1):3-10. doi: 10.5301/hipint.5000556. PMID 28983887
- [Background] Gausden EB, Qudsi R, Boone MD, O'Gara B, Ruzbarsky JJ, Lorich DG. Tranexamic Acid in Orthopaedic Trauma Surgery: A Meta-Analysis. J Orthop Trauma. 2017 Oct;31(10):513-519. doi: 10.1097/BOT.0000000000000913. PMID 28938281
- [Background] Franchini M, Mengoli C, Marietta M, Marano G, Vaglio S, Pupella S, Mannucci PM, Liumbruno GM. Safety of intravenous tranexamic acid in patients undergoing majororthopaedic surgery: a meta-analysis of randomised controlled trials. Blood Transfus. 2018 Jan;16(1):36-43. doi: 10.2450//2017.0219-17. PMID 29337665
- [Background] Hooda B, Chouhan RS, Rath GP, Bithal PK, Suri A, Lamsal R. Effect of tranexamic acid on intraoperative blood loss and transfusion requirements in patients undergoing excision of intracranial meningioma. J Clin Neurosci. 2017 Jul;41:132-138. doi: 10.1016/j.jocn.2017.02.053. Epub 2017 Mar 7. PMID 28283245
- [Background] Franchini M, Mengoli C, Cruciani M, Bergamini V, Presti F, Marano G, Pupella S, Vaglio S, Masiello F, Veropalumbo E, Piccinini V, Pati I, Liumbruno GM. Safety and efficacy of tranexamic acid for prevention of obstetric haemorrhage: an updated systematic review and meta-analysis. Blood Transfus. 2018 Jul;16(4):329-337. doi: 10.2450/2018.0026-18. Epub 2018 Apr 3. PMID 29757132
- [Background] Ali Algadiem E, Aleisa AA, Alsubaie HI, Buhlaiqah NR, Algadeeb JB, Alsneini HA. Blood Loss Estimation Using Gauze Visual Analogue. Trauma Mon. 2016 May 3;21(2):e34131. doi: 10.5812/traumamon.34131. eCollection 2016 May. PMID 27626017
- [Background] Goobie SM, Zurakowski D, Glotzbecker MP, McCann ME, Hedequist D, Brustowicz RM, Sethna NF, Karlin LI, Emans JB, Hresko MT. Tranexamic Acid Is Efficacious at Decreasing the Rate of Blood Loss in Adolescent Scoliosis Surgery: A Randomized Placebo-Controlled Trial. J Bone Joint Surg Am. 2018 Dec 5;100(23):2024-2032. doi: 10.2106/JBJS.18.00314. PMID 30516625
- [Background] Cuff DJ, Simon P, Gorman RA 2nd. Randomized prospective evaluation of the use of tranexamic acid and effects on blood loss for proximal humeral fracture surgery. J Shoulder Elbow Surg. 2020 Aug;29(8):1627-1632. doi: 10.1016/j.jse.2020.04.016. Epub 2020 Jun 9. PMID 32713466
- [Background] Yang YY, Qin H, Zheng X, Hu B, Zhang M, Ma T. Administration of Tranexamic Acid in Proximal Humeral Fractures. Indian J Orthop. 2020 May 11;54(Suppl 2):277-282. doi: 10.1007/s43465-020-00128-0. eCollection 2020 Dec. PMID 33194102